CLINICAL TRIAL: NCT04143815
Title: PhaseII, Randomized, Double-blind, Placebo Controlled, Multi-center, Dose-ranging and Open Label Extension Clinical Trial to Evaluate the Efficacy and Safety of MBA-P01 in Treatment of Moderate to Severe Glabellar Lines
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of MBA-P01 in Treatment of Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT14-AU18GBL208
Record Dates: First submitted 2019-10-28; First posted 2019-10-29 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MBA-P01 30U (Experimental): Experimental group, Dose: 30U
  Interventions: Drug: MBA-P01 (Botulinum toxin A)
- MBA-P01 20U (Experimental): Experimental group, Dose: 20U
  Interventions: Drug: MBA-P01 (Botulinum toxin A)
- MBA-P01 10U (Experimental): Experimental group, Dose: 10U
  Interventions: Drug: MBA-P01 (Botulinum toxin A)
- Placebo (Placebo Comparator): Placebo group, Normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBA-P01 (Botulinum toxin A) — Intramuscular injection, dose varies by groups
  Arms: MBA-P01 10U; MBA-P01 20U; MBA-P01 30U
Drug: Placebo — Intramuscular injection
  Arms: Placebo

SUMMARY:
This study will determine the effect of MBA-P01 in subjects with glabellar lines at a range of doses compared with placebo.

This study includes two treatment period; 1) Dose-ranging period, Day0 to 16weeks and 2) Open-label extension period, 16 weeks to 52.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age
* Bilaterally symmetrical moderate to severe GL at maximum frown as assessed by both investigator and subject using FWS

Exclusion Criteria:

* History of facial nerve paralysis
* Any eyebrow or eyelied ptosis as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Facial Wrinkle Scale(FWS) change | 4 weeks
  Proportion of subjects achieving at least a 2-grade decrease from baseline in score of Facial Wrinkle Scale (FWS) (0:none to 3: severe) of Glabellar line at maximum frown

CONTACTS AND LOCATIONS:
Locations (1):
- Maroubra MEdical Centre, Maroubra, New South Wales, Australia